CLINICAL TRIAL: NCT03130790
Title: A Two-Part Phase 2/ 3 Multicentre, Double-Blind, Randomized, Placebo Controlled Study of Varlitinib Plus mFOLFOX6 Verses Placebo Plus mFOLFOX6 In Subjects With HER1/ HER2 Co Expressing Advanced or Metastatic Gastric Cancer Without Prior Exposure to Systemic Therapy
Brief Title: Varlitinib in Combination With mFOLFOX6 for Advanced or Metastatic Gastric Cancer (First Line)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ASLAN Pharmaceuticals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASLAN001-012
Record Dates: First submitted 2017-04-16; First posted 2017-04-26 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — ARRY-334543

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Varlititib+mFOLFOX6 (Experimental)
  Interventions: Drug: Varlitinib; Drug: mFOLFOX6
- Placebo+mFOLFOX6 (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: mFOLFOX6

INTERVENTIONS:
Drug: Varlitinib — 300mg, oral tablets, twice daily for 2 weeks. Number of cycles: until disease progression, unacceptable toxicity, withdrawal of consent, or death.
  Other Names: ASLAN001; ARRY-334543; SPS4370; QBT01
  Arms: Varlititib+mFOLFOX6
Drug: mFOLFOX6 — concurrent oxaliplatin 85 mg/m2 and leucovorin 400 mg/m2 IV in 500 ml 5% dextrose water (D5W) over 120 minutes on Day 1; then 5 Fluorouracil bolus 400 mg/m2 IV on Day 1 followed by continuous infusion 2400 mg/ m2 over 46 hours starting on Day 1) every 2 weeks. Number of cycles: until disease progression, unacceptable toxicity, withdrawal of consent, or death.
  Arms: Varlititib+mFOLFOX6
Drug: Placebo — oral tablets, twice daily for 2 weeks. Number of cycles: until disease progression, unacceptable toxicity, withdrawal of consent, or death.
  Arms: Placebo+mFOLFOX6
Drug: mFOLFOX6 — concurrent oxaliplatin 85 mg/m2 and leucovorin 400 mg/m2 IV in 500 ml 5% dextrose water (D5W) over 120 minutes on Day 1; then 5 Fluorouracil bolus 400 mg/m2 IV on Day 1 followed by continuous infusion 2400 mg/ m2 over 46 hours starting on Day 1) every 2 weeks. Number of cycles: until disease progression, unacceptable toxicity, withdrawal of consent, or death.
  Arms: Placebo+mFOLFOX6

SUMMARY:
This protocol for Varlitinib is developed for the treatment of Gastric Cancer. Varlitinib (also known as ASLAN001) is a small-molecule, adenosine triphosphate competitive inhibitor of the tyrosine kinases - epidermal growth factor receptor (EGFR), human epidermal growth factor receptor (HER)2, and HER4. Varlitinib may be beneficial to subjects with cancer by simultaneous inhibition of these receptors. The purpose of this study is to determine the safety and efficacy of Varlitinib in combination with mFOLFOX6 for the treatment of Gastric Cancer. Treatment groups are Varlitinib+mFOLFOX6 and Placebo+mFOLFOX6.

DETAILED DESCRIPTION:
Phase 2 is planned to recruit approximately 50 or more eligible subjects in order to obtain data from 40 evaluable patients. Anticipated completion date in Dec 2018. Recruitment completed.

Phase 3 is planned to recruit 350 patients. Anticipated completion date in Dec 2022. Not yet recruiting.

ELIGIBILITY:
Inclusion Criteria - Phase 2 Part

1. Subjects of respective country's legal age or older at the time of written informed consent.
2. Subjects with histologically confirmed inoperable locally advanced, recurrent, or metastatic adenocarcinoma of the stomach or GEJ cancers may include Siewert Class I, II, or III types.
3. Mandatory provision of an unstained, archived tumor tissue sample in a quantity sufficient to allow for local lab analysis of HER1 and HER2 expression status. If archived tumor tissue is not available, subject must agree to undergo fresh core biopsy to obtain adequate tumor tissue
4. Subjects with tumors with IHC evidence of expression of HER1 (at level of + or ++ or +++) and HER-2 (at level of +, or ++) using standard criteria in the local lab. Subjects with HER-2 over expression at level of +++ determined by IHC and subject confirmed HER2 2+ by IHC with HER2 gene amplification confirmed by FISH but has contradiction to trastuzumab*.

   *For details of contraindication related to trastuzumab, refer to package insert or US treatment guideline.
5. Have radiographically measurable disease as defined by RECIST v1.1
6. Subjects with Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
7. Estimated life expectancy of more than 4 months
8. Able to swallow and retain oral medication
9. Subject with adequate organ and hematological function:

   d) Hematological function, as follows: i. Absolute neutrophil count (ANC) ≥1.5 x 109/L ii. Platelet count ≥ 100 x 109/L iii. HgB≥9 g/dL (packed red cell blood transfusions are not allowed within one week prior to baseline hematology profile).

   e) Renal functions, as follows: i. Serum creatinine ≤1.5x upper limit of normal (ULN) or estimated glomerular filtration rate (eGFR)> 60 mL/min/1.73m2 f) Hepatic function, as follows: i. Total bilirubin ≤1.5 x ULN ii. AST and ALT ≤2.5 x ULN (or ≤5 x ULN in subjects with liver metastasis) iii. Albumin ≥25 g/L
10. Negative serum human chorionic gonadotropin (HCG)/ or urine pregnancy test within 7 days prior to randomization for premenopausal women of reproductive capacity and for women 12 months after menopause
11. Willingness to use highly effective birth control method (failure rate <1%) while on study.

Inclusion Criteria - Phase 3 Part

1. Subjects of respective country's legal age or older at the time of written informed consent.
2. Subjects with histologically confirmed inoperable locally advanced, recurrent, or metastatic adenocarcinoma of the stomach or GEJ cancers may include Siewert Class I, II, or III types.
3. Mandatory provision of an unstained, archived tumor tissue sample in a quantity sufficient to allow for local lab analysis of HER1 and HER2 expression status. If archived tumor tissue is not available, subject must agree to undergo fresh core biopsy to obtain adequate tumor tissue.
4. Subjects with tumors with IHC evidence of expression of HER1 (at level of + or ++ or +++) and HER-2 (at level of +, or ++) using standard criteria in the local lab. Subjects with HER-2 over expression at level of +++ determined by IHC and subject confirmed HER2 2+ by IHC with HER2 gene amplification confirmed by FISH but has contradiction to trastuzumab*.
5. Note: *For details of contraindication related to trastuzumab, refer to package insert or US treatment guideline
6. Subjects with ECOG performance status of 0 to 1
7. Able to swallow and retain oral medication
8. Subject with adequate organ and hematological function:

   a) Hematological function, as follows: i. Absolute neutrophil count (ANC) ≥1.5 x 109/L ii. Platelet count ≥100 x 109/L iii. HgB≥9 g/dL (packed red cell blood transfusions are not allowed within one week prior to baseline hematology profile).

   b) Renal functions, as follows: i. Serum creatinine ≤ 1.5x ULN or eGFR> 60 mL/min/1.73m2 c) Hepatic function, as follows: i. Total bilirubin ≤1.5 x ULN ii. AST and ALT ≤2.5 x ULN (or ≤5 x ULN in subjects with liver metastasis) iii. Albumin ≥25 g/L
9. Negative serum human chorionic gonadotropin (HCG)/ or urine pregnancy test within 7 days prior to randomization for premenopausal women of reproductive capacity and for women 12 months after menopause
10. Willingness to use highly effective birth control method (failure rate <1%) while on study.

Exclusion Criteria:

1. Subject with HER-2 over expression at level of +++ determined by IHC or subject confirmed HER2 2+ by IHC with HER2 gene amplification confirmed by Fluorescence in situ hybridization (FISH) in the central lab.
2. Prior systemic anti-cancer treatment for inoperable locally advanced, recurrent, or metastatic adenocarcinoma of the stomach or GEJ. However, previous neo adjuvant chemotherapy is allowed if subject has progression of disease more than 6 months after neoadjuvant treatment.
3. Subjects have undergone major surgery within 28 days prior to randomization
4. Subject with brain lesion, known brain metastases (unless previously treated and well controlled for a period of at least 4weeks).
5. Subject with malabsorption syndrome, diseases significantly affecting gastrointestinal function, extensive resection of the stomach or small bowel, or difficulty in swallowing and retaining oral medications.
6. Subjects with an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, New York heart Association class III or IV congestive heart failure, unstable angina pectoris, clinically significant cardiac arrhythmia, diabetes, hypertension, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Subjects with any history of other malignancy unless in remission for more than 1 year. (Nonmelanoma skin carcinoma and carcinoma-in-site of uterine cervix treated with curative intent is not exclusionary).
8. Female subjects who are pregnant or breast feeding.
9. Subjects who were previously treated with varlitinib.
10. Subjects who took other investigational drugs and/or used investigational medical devices or have undergone major surgery within 28 days before initiating varlitinib therapy.
11. Are currently on or have received anti-cancer therapy, radiation or local treatment within the past 28 days
12. Subject with unresolved or unstable serious toxicity (≥ CTCAE 4.03 Grade 2) from prior administration of another investigational drug and/or prior cancer treatment(excluding hair loss)
13. Subjects with a known history of human immunodeficiency virus (HIV), decompensated cirrhosis, hepatitis B infection with hepatitis B virus DNA exceeding 2000 IU/mL or hepatitis C (treatment naïve or after treatment without sustained virologic response).
14. Known history of drug addiction within the past 1 year.
15. Subjects who need continuous treatment with proton pump inhibitors during the study period.
16. Any history or presence of clinically significant cardiovascular, respiratory, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic or psychiatric disease or any other condition which in the opinion of the Investigator could jeopardize the safety of the subject or the validity of the study results.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline in tumor size at Week 12 - Phase 2 part | At baseline and every 6 weeks for 24 weeks, after which reduced to once every 12 weeks until progression (up to approximately 3 months)
  Phase 2 part: Percentage change in tumour size defined as the percentage change from baseline in the sum of longest diameters of target lesions as assessed by ICR and defined by the RECIST v1.1 criteria
Overall Survival (OS) - Phase 3 part | When 247 OS events have occured. 247 OS is estimated to occur after approximately 45 months
  Phase 3 part: Overall Survival (OS) defined as the time from randomization until death by any cause. Any subject not known to have died at the time of the analysis will be censored based on the last recorded date on which the subject was known to be alive.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) - Phase 2 part | At baseline and every 6 weeks for 24 weeks, after which reduced to once every 12 weeks until progression (up to approximately 12 months)
  Phase 2 part: Objective Response Rate (ORR) defined as the proportion of subjects with a best objective response (BOR) of complete response (CR) or partial response (PR), as defined by the RECIST v1.1 criteria.
Progression-free survival (PFS) - Phase 2 part | At baseline and every 6 weeks for 24 weeks, after which reduced to once every 12 weeks until progression (up to approximately 12 months)
  Phase 2 part: Progression-free survival (PFS) defined as the time from randomization until the date of objective disease progression or death (by any cause in the absence of disease progression), whichever comes first. Progression is defined in accordance with the RECIST v1.1 criteria.
Time to response (TTR) - Phase 2 part | At baseline and every 6 weeks for 24 weeks, after which reduced to once every 12 weeks until progression (up to approximately 12 months)
  Phase 2 part: Time to response (TTR) defined as the time between date of randomization and first documented response (CR or PR), in the subset of subjects classified as responders in the assessment of ORR.
Duration of Response (DoR) - Phase 2 part | At baseline and every 6 weeks for 24 weeks, after which reduced to once every 12 weeks until progression (up to approximately 12 months)
  Phase 2 part: Duration of Response (DoR) defined as the time, in days, from the first recorded achievement of a response (PR or above) until time of objective disease progression in the subset of subjects classified as responders in the assessment of ORR.
Disease Control Rate (DCR) - Phase 2 part | At baseline and every 6 weeks for 24 weeks, after which reduced to once every 12 weeks until progression (up to approximately 12 months)
  Phase 2 part: Disease Control Rate (DCR) defined as the proportion of subjects with a (BOR of CR or PR, or SD maintained for a minimum of twelve weeks (-5 days) from randomization, as defined by the RECIST v1.1 criteria.
Overall Survival (OS) - Phase 2 part | From randomization to end of study (Last subject last visit (LSLV)) (up to approximately 24 months)
  Phase 2 part: Overall Survival (OS) defined as the time from randomization until death by any cause. Any subject not known to have died at the time of the analysis will be censored based on the last recorded date on which the subject was known to be alive.
Pharmacokinetic: area under the plasma concentration time curve (AUC) from 0 to 6 hours (AUC0-6) - Phase 2 part | Pharmacokinetic measurements will be taken on pre-dose, 1, 3, and 6 hours post dose on Day 1 and on Day 15
  Phase 2 part: Pharmacokinetic of Varlitinib
Pharmacokinetic: maximum observed plasma concentration (Cmax) - Phase 2 part | Pharmacokinetic measurements will be taken on pre-dose, 1, 3, and 6 hours post dose on Day 1 and on Day 15
  Phase 2 part: Pharmacokinetic of Varlitinib
Pharmacokinetic: time to Cmax (tmax) - Phase 2 part | Pharmacokinetic measurements will be taken on pre-dose, 1, 3, and 6 hours post dose on Day 1 and on Day 15
  Phase 2 part: Pharmacokinetic of Varlitinib
Pharmacokinetic: accumulation ratio for AUC (Rac AUC0-6) - Phase 2 part | Pharmacokinetic measurements will be taken on pre-dose, 1, 3, and 6 hours post dose on Day 1 and on Day 15
  Phase 2 part: Pharmacokinetic of Varlitinib
Pharmacokinetic: accumulation ratio for Cmax (Rac Cmax) - Phase 2 part | Pharmacokinetic measurements will be taken on pre-dose, 1, 3, and 6 hours post dose on Day 1 and on Day 15
  Phase 2 part: Pharmacokinetic of Varlitinib
Objective Response Rate (ORR) - Phase 3 part | When 247 Overall Survival (OS) events have occured (up to approximately 45 months)
  Phase 3 part: Objective Response Rate (ORR) defined as the proportion of subjects with a best objective response (BOR) of complete response (CR) or partial response (PR), as defined by the RECIST v1.1 criteria.
Progression-free survival (PFS) - Phase 3 part | When 247 Overall Survival (OS) events have occured (up to approximately 45 months)
  Phase 3 part: Progression-free survival (PFS) defined as the time from randomization until the date of objective disease progression or death (by any cause in the absence of disease progression), whichever comes first. Progression is defined in accordance with the RECIST v1.1 criteria.
Time to response (TTR) - Phase 3 part | When 247 Overall Survival (OS) events have occured (up to approximately 45 months)
  Phase 3 part: Time to response (TTR) defined as the time between date of randomization and first documented response (CR or PR), in the subset of subjects classified as responders in the assessment of ORR.
Duration of Response (DoR) - Phase 3 part | When 247 Overall Survival (OS) events have occured (up to approximately 45 months)
  Phase 3 part: Duration of Response (DoR) defined as the time, in days, from the first recorded achievement of a response (PR or above) until time of objective disease progression in the subset of subjects classified as responders in the assessment of ORR.
Disease Control Rate (DCR) - Phase 3 part | When 247 Overall Survival (OS) events have occured (up to approximately 45 months)
  Phase 3 part: Disease Control Rate (DCR) defined as the proportion of subjects with a (BOR of CR or PR, or SD maintained for a minimum of twelve weeks (-5 days) from randomization, as defined by the RECIST v1.1 criteria.
Incidence of Adverse Events (AEs) - Phase 3 part | When 247 Overall Survival (OS) events have occured (up to approximately 45 months)
  Phase 3 part: Incidence of AEs, categorized in accordance to CTCAE 4.03 and changes from baseline in safety parameters (including vital signs, ECG parameters, clinical laboratory tests)
Health-related quality of life (QoL) - Phase 3 part | When 247 OS events have occured. 247 OS is estimated to occur after approximately 45 months
  QLQ-C30 and EORTC QLQ-STO22 questionnaire
European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Core 30 items (EORTC QLQ-C30) measuring patients general cancer symptoms and functioning - Phase 3 part | When 247 OS events have occured. 247 OS is estimated to occur after approximately 45 months
  Phase 3 part: To assess on disease-related symptoms and health-related quality of life (QoL) of gastric cancer patients
European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Gastric Cancer 22 items (EORTC QLQ STO22) measuring patients general cancer symptoms and functioning - Phase 3 part | When 247 OS events have occured. 247 OS is estimated to occur after approximately 45 months
  Phase 3 part: To assess on disease-related symptoms and health-related quality of life (QoL) of gastric cancer patients

CONTACTS AND LOCATIONS:
Locations (16):
- 2 Sites, Tallinn, Estonia
- 1 Site, Hong Kong, Hong Kong
- Lithuania (2):
  - 2 Sites, Kaunas
  - 1 Site, Vilnius
- 2 Sites, Kuala Lumpur, Malaysia
- 1 Site, Singapore, Singapore
- South Korea (5):
  - 2 Sites, Daegu
  - 1 Site, Incheon
  - 1 Site, Jeongnam
  - 11 Sites, Seoul
  - 2 Sites, Suwon
- Taiwan (3):
  - 1 Site, Kaohsiung City
  - 1 Site, Taichung
  - 1 Site, Taipei
- Thailand (2):
  - 1 Site, Khon Kaen
  - 1 Site, Pathum Thani

IPD SHARING:
Plan to Share IPD: No